CLINICAL TRIAL: NCT06531395
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of Abiprubart in Participants With Sjögren's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Abiprubart in Participants With Sjögren's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to strategic business decision.
Sponsor: Kiniksa Pharmaceuticals International, plc (Industry)
Collaborators: Kiniksa Pharmaceuticals, GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPL-404-C221; 2024-512986-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Sjögrens Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Abiprubart 400mg SC q2wk (Experimental): Part A: Loading dose of abiprubart 800 mg subcutaneous (SC) followed by abiprubart 400 mg SC every 2 weeks (q2wk) through Week 22.
  Part B: Abiprubart 400 mg SC q2wk: abiprubart 400 mg SC q2wk up to and including Week 46.
  Interventions: Drug: Abiprubart
- Abiprubart 400mg SC q4wk (Experimental): Part A: Loading dose of abiprubart 800 mg SC followed by abiprubart 400 mg SC q2wk through Week 22 which will alternately administer placebo or abiprubart to provide active drug every 4 weeks (q4wk) while maintaining treatment concealment.
  Part B: Abiprubart 400 mg SC q4wk: abiprubart 400 mg SC q2wk up to and including Week 46 which will alternately administer placebo or abiprubart to provide active drug q4wk while maintaining treatment concealment.
  Interventions: Drug: Abiprubart; Drug: Placebo
- Placebo (Placebo Comparator): Part A: A matched volume placebo loading dose followed by placebo SC injections q2wk through Week 22.
  Part B: Participants assigned to placebo in Part A will transition to active abiprubart treatment, according to randomized assignment, with either abiprubart 400 mg SC q2wk or abiprubart 400 mg SC q4wk.
  Interventions: Drug: Abiprubart; Drug: Placebo

INTERVENTIONS:
Drug: Abiprubart — humanized monoclonal antibody
  Other Names: KPL-404
Drug: Placebo — sterile preservative-free solution
  Arms: Abiprubart 400mg SC q4wk; Placebo

SUMMARY:
Primary objective of the study is to evaluate the effect of abiprubart on an established systemic disease activity measure for Sjögren's Disease.

DETAILED DESCRIPTION:
This is a 56-week (24-week randomized double-blind period, 24-week active treatment period, and 8-week safety follow-up period) multicenter, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the efficacy and safety of abiprubart in participants with Sjögren's Disease with moderate or high systemic disease activity according to the European League Against Rheumatism (EULAR) Sjögren's Syndrome Disease Activity Index (ESSDAI). The objectives of the study are to evaluate efficacy, safety, pharmacokinetics (PK), and pharmacodynamics (PD) of abiprubart compared with placebo across the estimated therapeutic range using different dosing regimens of abiprubart.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of Sjögren's Disease according to 2016 American College or Rheumatology (ACR)-EULAR Classification Criteria.
* Has ESSDAI value ≥ 5, counting only the biological, hematological, articular, cutaneous, glandular, lymphadenopathy, and constitutional organ domains at Screening.
* Is seropositive at Screening for anti-Sjögren's-syndrome-related antigen A autoantibodies (SSA) antibodies tested at a central laboratory.
* Has stimulated whole salivary flow rate at Screening of ≥ 0.05 mL/min
* Weighs at least 40 kg and no more than 150 kg and has a body mass index (BMI) within the range of 18-40 kg/m2.

Exclusion Criteria:

* Prior exposure to any other anti-CD40/CD154 agent.
* Diagnosis of Sjögren's Disease overlap syndromes where another autoimmune rheumatic disease constitutes the principal illness, including fibromyalgia with currently active, inadequately controlled symptoms.
* Has received cataract surgery, Lasik, or other ophthalmologic surgery procedure (e.g., lachrymal plug) in the 6 months prior to Screening.
* Injectable corticosteroids (including intra-articular) within 8 weeks prior to randomization.
* Has started, stopped or adjusted dose/regimen of medications for treatment of, or known to cause dry mouth/eyes within the 30 days prior to screening or is anticipating change to these treatment regimens during the study.
* Has history of immunodeficiency (e.g., immune disorders or disorders that result in decreased immunity), including human immunodeficiency virus (HIV).
* History of thromboembolic event or a significant risk of future thromboembolic events.
* Has a known high risk of infection; Has a history of chronic or recurrent infectious disease; Has any known or suspected active infection, or has had a serious infection requiring hospitalization, or has been treated with IV/IM antibiotics for an infection within 8 weeks prior to first dose of study drug or treatment with oral antibiotics for an infection within 2 weeks prior to first dose of study drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in European League Against Rheumatism (EULAR) Sjögren's Syndrome Disease Activity Index (ESSDAI) at Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Proportion of Sjögren's Tool for Assessing Response (STAR) Responders (≥ 5 points) at Week 24 | Week 24
Proportion of STAR Responders (≥ 5 points) Over Time | Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 52, 56
Change From Baseline in Stimulated Salivary Flow Rate (mL/min) at Week 24 | Baseline, Week 24
Change From Baseline in Stimulated Salivary Flow Rate (mL/min) Over Time | Baseline, Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 52, 56
Change From Baseline in Unstimulated Salivary Flow Rate (mL/min) at Week 24 | Baseline, Week 24
Change From Baseline in Unstimulated Salivary Flow Rate (mL/min) Over Time | Baseline, Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 52, 56
Change From Baseline in EULAR Sjögren's Syndrome Disease Patient Reported Index (ESSPRI) at Week 24 | Baseline, Week 24
Change From Baseline in ESSPRI Over Time | Baseline, Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 52, 56
Change From Baseline in Schirmer's Test at Week 24 | Baseline, Week 24
Change From Baseline in Schirmer's Test Over Time | Baseline, Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 52, 56
Change From Baseline in Clinical EULAR Sjögren's Syndrome Disease Activity Index (clinESSDAI) at Week 24 | Baseline, Week 24
Change From Baseline in clinESSDAI Over Time | Baseline, Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 52, 56
Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) at Week 24 | Baseline, Week 24
Change From Baseline in FACIT-Fatigue Over Time | Baseline, Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 52, 56
Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D 5L) at Week 24 | Baseline, Week 24
Change From Baseline in EQ-5D 5L Over Time | Baseline, Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 52, 56

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Medvin Clinical Research, Menifee, California
  - BioSolutions Clinical Research Center, Poway, California
  - Medvin Clinical Research, Whittier, California
  - International Medical Research, Daytona Beach, Florida
  - Omega Research Debary, LLC, DeBary, Florida
  - Greater Chicago Specialty Physicians/ Clinical Investigation Specialists, Schaumburg, Illinois
  - Clinic of Robert Hozman, MD/Clinical Investigation Specialists, Inc., Skokie, Illinois
  - Springfield Clinic Rheumatology, Springfield, Illinois
  - Accurate Clinical Research, Inc, Lake Charles, Louisiana
  - Accellacare (Salisbury), Salisbury, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Arthritis and Rheumatology Research Institute, PLLC, Allen, Texas
  - Arthritis Care of Texas, Corpus Christi, Texas
  - Trinity Universal Research Associates, Inc., Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Arthritis & Osteoporosis Clinic, Waco, Texas

IPD SHARING:
Plan to Share IPD: No